CLINICAL TRIAL: NCT04801147
Title: Phase I Clinical Trial Of Immunotherapy With Autologous Tumor Lysate-Loaded Dendritic Cells In Patients With Newly Diagnosed Glioblastoma Multiforme (DENDR1)
Brief Title: Immunotherapy With Autologous Tumor Lysate-Loaded Dendritic Cells In Patients With Newly Diagnosed Glioblastoma Multiforme
Acronym: DENDR1
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DENDR1
Record Dates: First submitted 2021-03-09; First posted 2021-03-16 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-01

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: Phase I, 2-stage Simon design (Simon et al., 1997), single-centre, uncontrolled, open label, non-randomized study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy (Experimental): Autologous DC loaded with a autologous tumor lysate, in order to stimulate the immune response of the patient.
  Interventions: Biological: Dendritic Cells Vaccine

INTERVENTIONS:
Biological: Dendritic Cells Vaccine — Right after the surgical resection of the tumor, leukapheresis will be performed.
  At least 5x109 PBMC must be collected by leukapheresis, so as to make the whole immunotherapy schedule workable.
  Immunotherapy will follow radiochemotherapy and will comprise 4 vaccinations every second week (injections I, II, III, IV), 2 further monthly vaccinations (injections V, VI) and a final vaccination (injection VII) 2 months after the sixth one. Injections I, V, VI and VII will contain 10 million tumor lysate-loaded DC, while the others will be of 5 million cells only. In correspondence to the third vaccine injection (week 13), mTMZ will start.
  Vaccine doses will be injected in the forearm of the patient.

SUMMARY:
Rationale of the Study: Treatment for GBM currently consists of surgical resection of the tumour mass followed by radio- and chemotherapy ((1)Stupp et al., 2005). Nonetheless overall prognosis still remains bleak, recurrence is universal, and recurrent GBM patients clearly need innovative therapies. Dendritic cells (DC) immunotherapy could represent a well-tolerated, long-term tumour-specific treatment to kill all (residual) tumour cells which infiltrate in the adjacent areas of the brain. Preclinical investigations for the development of therapeutic vaccines against high grade gliomas, based on the use of DC loaded with a mixture of glioma-derived tumor have been carried out in rat as well as in mouse models, showing the capacity to generate a glioma-specific immune response. Mature DC loaded with autologous tumor lysate have been used also for the treatment of patients with recurrent malignant brain tumors; no major adverse events have been registered. Results about the use of immunotherapy for GBM patients are encouraging, but further studies are necessary to find out the most effective and safe combination of immunotherapy with radio- and chemotherapy after exeresis of the tumour mass.

Aim of the study. Primary objective of the study is to evaluate treatment tolerability and to get preliminary information about efficacy. Secondary objective is to evaluate the treatment effect on the immune response. Additional objective is to identify a possible correlation between methylation status of MGMT promoter and tumor response to treatment.

A two-stage Simon design ((2)Simon, 1989) will be considered for the study. Assuming as outcome measure the percentage of PFS12 patients and of clinical interest an increase to 42% (P1) of the historical control rate of 27% (P0) ((1)Stupp et al., 2005), the alternative hypothesis will be rejected at the end of the first stage if the PFS12 rate will be less than 8/24 treated patients (Fisher's exact test). In the second stage patients will be enrolled up to 76 overall. The null hypothesis will be rejected (a=0.05, b=0.2) if at least 27 subjects out of 76 are alive and progression free 12 months after the beginning of the treatment.

DETAILED DESCRIPTION:
Background and significance. The therapeutic program will include radical surgical resection of the tumor, followed by radiotherapy (fractionated local field irradiation in daily fractions of 2 Gy given 5 days per week, Monday through Friday for 6 weeks, for a total of 60 Gy) plus temozolomide (TMZ) chemotherapy (75 mg per square meter of body-surface area per day, 7 days per week from the first to the last day of radiotherapy). After a 4-week break, up to 6 cycles of maintenance TMZ (mTMZ) will be administered according to the standard 5-day (oral intake) schedule every 28 days. TMZ dose will be 150 mg per square meter for the first cycle and will be increased to 200 mg per square meter beginning with the second cycle, so long as there is no hematologic toxic effect. Immunotherapy will follow radiochemotherapy and will comprise 4 vaccinations every second week (injections I, II, III, IV), 2 further monthly vaccinations (injections V, VI) and a final vaccination (injection VII) 2 months after the sixth one. Injections I, V, VI and VII will contain 10 million tumor lysate-loaded DC, while the others will be of 5 million cells only. In correspondence to the third vaccine injection (week 13), mTMZ will start. On the basis of the patient clinical status, further vaccine boosts will be considered as appropriate addition at the standard vaccination cycle.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤70 years.
* Postoperative Karnofsky Performance Status ≥70.
* First diagnosis of GBM (World Health Organization [WHO] grade IV astrocytoma).
* Diagnosis confirmed by the reference histopathology.
* Residual tumor volume after resection <10 cc, confirmed by postoperative MRI assessment
* Total or subtotal resection of tumor mass, confirmed by assessment of the neurosurgeon and by postoperative radiological assessment.
* Amount of non-necrotic tissue for lysate preparation and DC loading ≥1 gr, stored at -80°C.
* Corticosteroids daily dose ≤4 mg during the 2 days prior to leukapheresis.
* Clinical indication for radiochemotherapy according to the Stupp protocol (Stupp et al., 2005).
* Life expectancy > 3 months.
* Informed consent

Exclusion Criteria:

* Pregnancy.
* Participation in other clinical trials with experimental drugs simultaneously or within 1 month before this trial entry.
* Presence of acute infection requiring active treatment.
* Mandatory treatment with corticosteroids or salicylates in anti-inflammatory dose.
* Presence of sub-ependymal diffusion of the tumor.
* Presence of multi-focal GBM lesions.
* Haematology: leukocytes < 3,000/μl, lymphocytes < 500/μl, neutrophils < 1,000/μl, hemoglobin <9 g/100 ml, thrombocytes < 100,000/μl one or two days prior to leukapheresis.
* Documented immune deficiency.
* Documented autoimmune disease.
* Positive serology for HIV, HBs antigen, HCV, TPHA.
* Allergies to any component of the DC vaccine.
* Known intolerance to TMZ.
* Other active malignancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2010-06-26 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Progression Free Survival | PFS12 is defined as the percentage of participants with PFS at 12 months from the date of surgery for newly diagnosed tumor to the first date of objectively determined progressive disease based on Response Assessment in Neuro-Oncology (RANO) criteria
  PFS12 is defined as the percentage of participants with PFS at 12 months from the date of surgery for newly diagnosed tumor to the first date of objectively determined progressive disease based on Response Assessment in Neuro-Oncology (RANO) criteria ((3)Wen et al JCO 2010) or death from any cause. It is assumed that PFS follows an exponential distribution. Estimation using Kaplan-Meier analysis.

SECONDARY OUTCOMES:
Incidence of Treatment-related Adverse Events | Tolerability will be monitored throughout study completion: during active treatment at least on vaccination-time points, and later an average of 2 months
  Tolerability will be assessed using CTCAE version 3.0 and recording incidence, severity and type of adverse events.
Evaluation of the treatment effect on the immune response | baseline (Leukapheresis)/ at each DC vaccine/every 2 months (from the end of DC vaccine)/ up through study competion, an avarage of 1 years.
  Immune response will be monitored throughout study completion: during active treatment at least on vaccination-time points, and later an average of 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Neuro-oncologia Molecolare, Milan, Italy

IPD SHARING:
Plan to Share IPD: No